CLINICAL TRIAL: NCT06492603
Title: Examination of Linea Alba Biomechanical and Viscoelastic Characteristics in Patients Diagnosed With Diastasis Recti Using Ultrasound
Brief Title: Examination of Biomechanical Characteristics of Linea Alba in Diastasis Recti Patients
Status: Not yet recruiting | Type: Observational
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Abouelyazeed Ali, Lecturer of Physical Therapy for Women's Health, South Valley University
Other Study IDs: Diastasis Recti
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2024-07

CONDITIONS: Separated Recti Abdominis
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- 20 Women in the Postpartum Diastasis Recti Group
  Interventions: Device: Ultrasonography; Device: The MyotonPRO Device
- 20 Women in the Control Group (Postpartum Without Diastasis Recti)
  Interventions: Device: Ultrasonography; Device: The MyotonPRO Device

INTERVENTIONS:
Device: Ultrasonography — Ultrasound is an assessment device that uses high-energy sound waves to look at either superficial tissues like linea alba and/or organs inside the body. The sound waves make echoes that form pictures of the tissues and organs on a computer screen (sonogram).
Device: The MyotonPRO Device — The MyotonPro is a portable device for measuring biomechanical and viscoelastic properties in superficial soft tissues

SUMMARY:
Diastasis recti is an increased distance between the rectus abdominis muscles at the midline caused by weakness in the anterior abdominal wall.

DETAILED DESCRIPTION:
Most healthcare providers agree that in diastasis rectus abdominis there is a weakness, thinning, and widening of the linea alba and weakness of the associated abdominal musculature.

Ultrasonography is regarded as the most accurate method for measuring the IRD and its results are consistent with the data derived from palpation, calipers, and intraoperative measurements.

The MyotonPRO Device is used for the non-invasive measurement of Device is for the non-invasive measurement of biomechanical and viscoelastic properties of superficial soft biological tissues. Skeletal muscles or tendons can be measured at different regions, at full rest or in contraction.

This study aims to assess the biomechanical and viscoelastic properties of the Linea Alba in patients who are diagnosed with diastasis rectus abdominis by ultrasonography.

ELIGIBILITY:
Inclusion Criteria:

* Postpartum Mothers who delivered by a cesarean section.
* Postpartum Mothers with a BMI below 30 or a Waist-hip ratio below 1.
* Postpartum Mothers above 18 years old and those below 40 years old.

Exclusion Criteria:

* Postpartum Mothers who delivered by a vaginal delivery.
* Postpartum Mothers who had hernias in the abdominal region or laparotomy.
* Postpartum Mothers with a BMI over 30 or a Waist-hip ratio over 1.
* Postpartum Mothers below 18 years old and those above 40 years old.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study examines the Biomechanical and Viscoelastic Characteristics of Diastasis Rectus Abdominis in Postpartum Women
Study Population: 40 post-Cesarean women who are diagnosed with or without diastasis rectus abdominis. They will be selected from the teaching Hospitals of South Valley University.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-07-20 (Estimated); Primary Completion 2025-11-20 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Linea Alba Stiffness | Assessment will be done at the 7th day postpartum and at the end of the 6th week postpartum
  It is a Biomechanical Characteristic of the Linea Alba
Linea Alba Elasticity | Assessment will be done at the 7th day postpartum and at the end of the 6th week postpartum
  It is a Biomechanical Characteristic of the Linea Alba
Linea Alba Creep | Assessment will be done at the 7th day postpartum and at the end of the 6th week postpartum
  It is a Viscoelastic Characteristic of the Linea Alba

IPD SHARING:
Plan to Share IPD: No